CLINICAL TRIAL: NCT00657527
Title: An 8-Week Randomized Double Blind Placebo Controlled Multicenter Trial to Evaluate the Effects of Rosuvastatin 40mg on Myocardial Ischemia in Subjects With Coronary Artery Disease.
Brief Title: Evaluation of Effects of Rosuvastatin 40mg on Myocardial Ischemia in Subjects With Coronary Artery Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Elisabeth Björk, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4522IL/0043; D3560C00043
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2009-03-16 (Estimated); Status verified 2009-03

CONDITIONS: Myocardial Ischaemia; Coronary Artery Disease
Keywords: Crestor; Rosuvastatin; Cholesterol; Coronary artery disease; Myocardial ischaemia.
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rosuvastatin
  Interventions: Drug: Rosuvastatin
- 2 (No Intervention): Diet
  Interventions: Behavioral: Cholesterol lowering diet

INTERVENTIONS:
Drug: Rosuvastatin
  Other Names: Crestor
  Arms: 1
Behavioral: Cholesterol lowering diet
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether treatment with 40mg of Rosuvastatin for 8 weeks will reduce the number of episodes of myocardial ischaemia suffered in subjects with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Coronary arterial disease
* Suffering ischaemic episodes/exercise induced ischaemia
* Not taking any cholesterol lowering medication

Exclusion Criteria:

* Unstable angina or heart attack less than one month before trial entry
* Coronary arterial surgery as defined by protocol
* Uncontrolled hypertension, diabetes, hypothyroidism or laboratory values as defined by the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2001-12; Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Number of episodes of myocardial ischaemia as assessed by ambulatory electrocardiographic monitoring. | 8 weekly

SECONDARY OUTCOMES:
Change in duration of ischemic episodes | 8 weekly
Safety | 8 weekly
Several laboratory parameters as detailed in the protocol | 8 weekly

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cressman, DO, Study Director — AstraZeneca; Russell Esterline, Study Chair — AstraZeneca